CLINICAL TRIAL: NCT05057039
Title: The Study of Gut Microbiota in Hypertensive Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Taipei Medical University (Other)
Collaborators: Cathay General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CGH-P110063
Record Dates: First submitted 2021-09-09; First posted 2021-09-27 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-01

CONDITIONS: Hypertension; Gut Microbiota; Diet
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hypertensive group: SBP >=140mmHg, DBP >=90mmHg, or use of antihypertensive drug
- normotensive group: SBP <=140mmHg and DBP <=90mmHg without use of antihypertensive drug

SUMMARY:
Recent animal and human studies have found the relationship between the composition of the gut microbiota and hypertension, but some studies did not have a detailed evaluation of the diet content, which could be an important effect on gut microbiota. Moreover, most of these studies were finished in Western countries, in which the dietary patterns were significantly different from those in Chinese regions. This study intends to establish Taiwanese local data to explore the differences in the composition of gut microbiota among hypertensive patients and normotensive subjects.

DETAILED DESCRIPTION:
The investigators plan to enroll total 70 hypertensive and normotensive cases from the elderly health examination in Cathay General Hospital, who are aged from 65 to 80 years. Body mass index and blood samples for biochemical analysis such as blood sugar and cholesterol levels are taken, and fecal samples are collected for analysis of gut microbiota, which is characterized by 16S ribosomal RNA gene sequencing. Besides, the diet and nutrients intake are recorded and calculated by licensed dietitian. Through the exploration of gut microbiota in hypertensive patients, the results can be the reference for clinical treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65~80 years old
2. People who join the Elderly Health Examination Program in Cathay General Hospital in 2021

Exclusion Criteria:

1. Antibiotics use within one month
2. Acute gastrointestinal illness within one week, such as vomiting and diarrhea
3. History of gastrointestinal surgery
4. History of inflammatory bowel disease
5. Chronic gastrointestinal disease under medication treatment
6. Cannot finish dietary record

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: People who join the Elderly Health Examination Program in Cathay General Hospital in 2021
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The difference of gut microbiota composition between the two groups | immediately after the enrollment completes
  The differential OTUs (operational taxonomic units) between the two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University, Taipei, Taiwan